CLINICAL TRIAL: NCT06017856
Title: The Impact of Physical Exercise and Nutrition on Functional Gastrointestinal Disorders in Obese Children
Brief Title: Physical Exercise and Nutrition in Functional Gastrointestinal Disorders in Obese Children
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, eyal zifman, Head of pediatric gastroeneterogy service, Meir Medical Center
Other Study IDs: MMC-22-0199
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Functional Gastrointestinal Disorders; Obesity, Childhood
Keywords: obese; overweight; abdominal pain; diarrhea
MeSH Terms: conditions — Gastrointestinal Diseases; Pediatric Obesity; Obesity; Overweight; Abdominal Pain; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese and overweight: Overweight and obese subjects, defined as body mass index (BMI) percentile ≥85%, participating the in life-style intervention program in the child sport center at Meir medical center
  Interventions: Other: Life style intervention program
- normal weight: normal weight subjects defined as body mass index (BMI) percentile <85%, with no other chronic conditions

INTERVENTIONS:
Other: Life style intervention program — Life style intervention program for the obese/overweight subjects conducted regardless of this study at the child sport and health center at Meir medical center
  Groups: obese and overweight

SUMMARY:
A prospective observational case-control study evaluating the effect of a weight loss intervention program on functional gastrointestinal disorders among overweight and obese children.

DETAILED DESCRIPTION:
The investigators intend to conduct a prospective observational case-control study of overweight and obese children, aged 6-18 years, followed in the child health and sport center at Meir medical center, Kfar-Saba, Israel.

Overweight and obese subjects, defined as body mass index (BMI) percentile ≥85%, will be offered to participate. Healthy subjects with normal BMI percentile from other pediatric outpatient clinics as well as relatives and friends of physicians from the pediatric division will be enrolled and serve as the control group.

Study visits will be at enrollment and after 3 and 6 months of participation in the intervention program. During the visits the investigators will collect anthropometric measurements (height, weight, BMI, total body fat). Participants (age 10y and above) or their parents (age 6-10y) will fill a validated questionnaire for diagnosis of FGID based on ROME IV criteria. The investigators will also collect data from exercise capability testing and quality of life questionnaires performed regularly (and irrespective of this study) during the intervention program.

The investigators will then compare between subjects who succeeded to those who failed in losing at least 5% of their initial body weight as well as to healthy controls with normal BMI percentile.

ELIGIBILITY:
Inclusion Criteria:

* obese / overweight children participating in the life style modification program at the child sport and health center

Exclusion Criteria:

* other known chronic non-functional gastrointestinal conditions (e.g. Celiac disease, inflammatory bowel disease)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: obese and overweight subjects patricipating in the life style modification program as well as healhy controls of normal weight
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of functional gastrointestinal disorder | 6 months
  The number of participants with a diagnosis of functional gastrointestinal disorder according to the Rome IV criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Zifman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No